CLINICAL TRIAL: NCT02594618
Title: Energy Metabolism and Cost of Physical Activities Using Whole Body Calorimeter
Status: Completed | Type: Observational
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Other Study IDs: 2014/00631
Record Dates: First submitted 2015-10-27; First posted 2015-11-03 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Energy Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to assess energy regulation of overfeeding and performing common household activities in young Chinese males using whole-body room calorimetry up to 10 hours.

DETAILED DESCRIPTION:
This study will require participants to stay in the room calorimeters for up to 5 hours on each of the 3 test sessions. The participants are to avoid intense physical activity/alcohol and to record their food intake for the day prior to test day. They will record their food intake for the day prior to test session 1 in a food diary (to be provided to them on the day of screening). Records will be used to ascertain participants' food intake patterns. They will report to Clinical Nutrition Research Centre (CNRC) in the morning after an overnight (10-12 hours) fast. Basic anthropometric measurements will be taken at the start of the test session before participants enter the room calorimeter. The room calorimeter is a 13.5 m3 chamber furnished with features to give an impression of a normal room with windows on three sides of the chamber for outside view and visual contact with researchers. It has a full sized foldaway bed, a fold-down writing table, an office chair, a built-in sink and mirror, a portable freeze-dry toilet bowl, a television, a telephone, computer network connection, an intercom system. During their stay in the room calorimeter, energy expenditure will be measured based on recorded oxygen consumption and carbon dioxide production over 10 hours. Participants are allowed to rest, sit and move freely, except sleep or exercise during their stay. On each of the 3 test sessions, the subjects will perform up to 4 common household activities (e.g. mopping floor, washing dishes, etc) 1 hour after consuming the light breakfast. On test session 1, the light breakfast consist of biscuits and a juice drink and will be provided to the participants after they have undergone assessment of metabolism at rest for approximately 45 minutes in the room calorimeter. On test session 2 and 3, the same light breakfast will be provided after approximately 15 minutes after they have entered the room calorimeter. During their 4-5 hours stay in the room calorimeter, they will simulate a particular household activity for up to 20 minutes and rest for 30 minutes before continuing with another household activity and so on for up to 4 different household activities at each of the test sessions.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Ethnic Chinese
* Age between 21 to 39 years
* Body mass 60 to 70 kg
* Body height 165 to 175 cm
* Normal resting blood pressure ~120/80 mmHg
* Normal fasting blood glucose level <5.5 mmol/L
* Do not train for or partake in competitive sports
* Do not have any major diseases
* Not on any prescribed medication
* Willing and able to consume all test meals
* Not allergic to any food ingredient found in all test meals

Ages: 21 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male healthy subjects who are of Chinese ethnicity
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
measuring energy cost of domestic physical activities using whole body calorimeter | 0 to 20 minutes
  Energy expenditure is measured for 20 minutes continuously throughout the domestic activity performed by the subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore